CLINICAL TRIAL: NCT03336424
Title: Prospective Randomized Controlled Trial Comparing the Non-invasive vs the Invasive Investigations in Multiple Sclerosis Patients With Urinary Disorders.
Brief Title: Urinary Disorders in Patients With Multiple Sclerosis: Invasive Vs Non-invasive Investigations.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FM292
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis; Urinary Bladder, Neurogenic; Urodynamics
Keywords: MS; Multiple sclerosis; urinary Bladder, Neurogenic; Urodynamics; Randomized controlled trial
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Parallel study, where group A receives non-invasive investigations and group B receives Invasive investigations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive investigations group (Experimental): Non-invasive investigations include: ultrasound, blood exam, urine analysis and culture, uroflowmetry
  Interventions: Diagnostic Test: Non-invasive investigations
- Invasive investigations group (Experimental): urodynamic study including: cystomanometry, pressure flow study, EMG
  Interventions: Diagnostic Test: Non-invasive investigations; Diagnostic Test: Invasive investigations

INTERVENTIONS:
Diagnostic Test: Non-invasive investigations — Ultrasound, blood tests, urine analysis and culture, uroflowmetry
Diagnostic Test: Invasive investigations — Cystomanometry, pressure flow study, EMG
  Arms: Invasive investigations group

SUMMARY:
The objective of the study is to describe the current status of MS patients with urinary disorders in Lebanon, and to demonstrate whether invasive investigations improve the management of these patients compared to an optimal non-invasive approach.

DETAILED DESCRIPTION:
All patients will be evaluated by an urologist, then randomized into 2 groups, the first group will benefit from non-invasive investigations and will be treated accordingly, the second group will benefit from an urodynamic assessment and will also be treated accordingly.

An evaluation will be made one month, 3 months and 6 months after the first visit.

ELIGIBILITY:
Inclusion Criteria:

* MS with urinary symptoms

Exclusion Criteria:

* BPH LUTS
* Bladder cancer
* prostate cancer
* urethral stenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
urinary symptoms | 6 months
  filling and voiding urinary symptoms (UBQMS: Urinary Bothersome Questionnaire in Multiple Sclerosis), Voising Score Ranges from 0 to 3 ( 3 being most severe bother), Filling score ranges from 0 to 3 ( 3 being most severe bother).
urinary quality of life | 6 months
  SF-QUALIVEEN: Short Form - health related quality of life questionnaire for urinary disorders in patients with neurological conditions. score ranges from 0 to 4 ( 4 being the worst quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Elie EL HELOU, MD, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No